CLINICAL TRIAL: NCT00850980
Title: Selective AV Nodal Vagal Stimulation For Reduction of the Ventricular Rate During Atrial Fibrillation
Status: Withdrawn | Type: Observational
Why Stopped: unable to recruit
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 08-766
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will enroll patients that are already in AF and in which open-heart surgical intervention has been scheduled. In these patients AVN-VNS will be delivered briefly (minutes) after the incision as a proof-of-concept therapy, with concomitant monitoring of the effects on the ventricular rate.

DETAILED DESCRIPTION:
Rate control during AF can be achieved by drugs (Ca++ blockers, digoxin, beta-blockers), or by AV nodal ablation. Drugs, as usual, have limitations, while the radical destruction of the AV node renders the patient permanently pacemaker-dependent.

In series of animal studies the investigators employed AVN-VNS delivered to the so-called AV nodal fat pad. Electrical stimulation of the fat pad resulted in release of neuromediator (acetylcholine) within the AV nodal domain. The investigators have demonstrated that this approach successfully and substantially slowed the ventricular rate during AF in both acute and chronic experiments without inflicting any damage on the AV node.

It is our hypothesis that temporary delivery of selective AVN-VNS in patients with AF will provide the benefits of reduced ventricular rate during the ongoing AF. The proposed study will be limited only to patients that are already in AF and in which open-heart surgical intervention has been scheduled. In these patients AVN-VNS will be delivered briefly (minutes) after the incision as a proof-of-concept therapy, with concomitant monitoring of the effects on the ventricular rate.

Based on the information obtained in this study, the investigators intend subsequently to test the AVN-VNS in a group of patients that develop AF post-operatively and remain in this status for several days after the surgery. A protocol for a separate study will be submitted if and when this becomes feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open heart surgery
* Able to give Informed Consent and
* Permanent/Persistent or currently in Atrial Fibrillation

Exclusion Criteria:

* Minimally invasive incisions
* Previous open heart surgery
* Bleeding diathesis
* Creatinine levels greater than 2.0 mg/dl
* Active Infections, i.e. endocarditis
* Implanted ICD
* Pregnancy and nursing
* Incompetence and/or other conditions, which do not allow the patient to understand the nature, significance and scope of the study
* Patients on drugs that have cholinesterase inhibitor activity (e.g., physostigmine-like substances).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery
  * Able to give Informed Consent and
  * Permanent/Persistent or currently in Atrial Fibrillation 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in ventricular rate from baseline measured at each amplitude | surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cleveland clinic research website — http://my.clevelandclinic.org/research